CLINICAL TRIAL: NCT00590031
Title: Preoperative Combined Modality Therapy for Esophageal Carcinoma: Cisplatin-Irinotecan Followed by Radiation Therapy With Concurrent Cisplatin and Irinotecan.
Brief Title: Phase II Trial of Preoperative Combined Modality Therapy for Esophageal Carcinoma: Cisplatin-Irinotecan Followed by Radiation Therapy With Concurrent Cisplatin and Irinotecan.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-045; IND 65889
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Results first posted 2016-01-25 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2015-12

CONDITIONS: Esophageal Carcinoma
Keywords: Esophageal Carcinoma; Cisplatin; Irinotecan; Radiation Therapy; 02-045
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Cisplatin; Irinotecan

ARMS (1):
- 1 (Experimental): External Beam Radiation Therapy, Cisplatin, Irinotecan
  Interventions: Drug: Cisplatin; Drug: Irinotecan; Radiation: External Beam Radiation Therapy

INTERVENTIONS:
Drug: Cisplatin — pts will receive weekly cisplatin 30mg/m2 after hydration on weeks 8,9,11 and 12
Drug: Irinotecan — Irinotecan will be given 65 mg/m2
Radiation: External Beam Radiation Therapy — will be delivered with multiple (>2) field techniques using mega-voltage radiation therapy. pts will receive 50.4 Gy and will be treated over a 6 week period.

SUMMARY:
Patients with surgically resectable T1N1M0 or T2-4N any M0 esophageal carcinoma will receive six weeks of induction chemotherapy with weekly irinotecan and cisplatin given weeks 1, 2, 4 and 5. Patients will then receive weekly irinotecan, cisplatin, and concurrent radiotherapy with chemotherapy given once weekly, weeks 8,9,11 and 12 during the six weeks of radiotherapy. Patients will be referred for surgery 4-8 weeks after completion of chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to sign the informed consent document.

Exclusion Criteria:

* Tis (in-situ carcinoma) and tumors determined to be TIN0 following endoscopy, endoscopic ultrasound, or CT scanning.
* Cervical esophageal tumors,
* Gastric cancers with minor involvement of the gastroesophageal junction or distal esophagus.
* Prior chemotherapy or radiation.
* Patients with evidence of metastatic disease are not eligible. This includes:
* Positive malignant cytology of the pleura, pericardium or peritoneum.
* Radiographic evidence of distant organ involvement including lung, liver, bone, or brain.
* Patients with involvement of non-regional lymph nodes including supraclavicular or celiac lymph node metastases.
* Biopsy proven tumor invasion of the tracheobronchial tree or presence of tracheoesophageal fistula. Recurrent laryngeal nerve or phrenic nerve paralysis,
* New York Heart Association Class III or 1V heart disease. Angina or myocardial infarction within the last 6 months, history of significant ventricular arrhythmia requiring medication with antiarrhythmics, or a history of a clinically significant conduction system abnormality.
* Severe co-morbid conditions including severe uncontrolled diabetes, uncontrolled hypertension, cerebral vascular disease, uncontrolled infection, or nonmalignant illness whose control may be jeopardized by the complications of this study treatment.
* Pregnant or lactating women are ineligible as the effect of the drugs used in this study on a fetus or newborn child are unknown. Premenopausal fertile females require a negative pregnancy test prior to study entry. Treatment may not begin until the results of the pregnancy tests are ascertained. Both sexes must use contraception while on this study.
* History of prior malignancy (other than basal cell/squamous carcinoma of the skin, in-situ cervical carcinoma, or superficial transitional cell bladder carcinoma) diagnosed and/or treated within three years of entrance into this study.
* Patients with known Gilbert's Disease.
* Clinically significant hearing loss.
* Serum calcium_>12 mg/dl.
* Patients with a history of seizure disorder who are receiving phenytoin, phenobarbital, or other antiepileptic medication.
* Patients who cannot fully comprehend the therapeutic implications of the protocol or comply with the requirements.
* Patients with any other concurrent medical or psychiatric condition or disease, which, in the investigator's judgment, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2002-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Ilson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Combined Modality Therapy for Esophageal Carcinoma: The trial will be a phase II, single institution trial of preoperative therapy with irinotecan, cisplatin, and concurrent radiotherapy in surgically resectable esophageal cancer. The primary endpoint is the pathologic complete response rate to preoperative therapy, and a sample size of 50 patients will characterize this response rate +/- 13% with 95% confidence. Secondary endpoints will include the toxicity of therapy, including surgical morbidity and mortality, the overall and disease-free survival, pattern of disease recurrence, and quality of life achieved during therapy, including relief of dysphagia.
Period: Overall Study
Arm/Group | Combined Modality Therapy for Esophageal Carcinoma
Started | 61
Completed | 55
Not Completed | 6
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — Metastatic Disease | 1
Not completed — Admin Hold | 1

BASELINE CHARACTERISTICS:
Arm/Group | Combined Modality Therapy for Esophageal Carcinoma
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 45
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response
Description: Pathological information will be available for all patients who receive surgery. If a patient is deemed unresectable based on clinical and radiological examination after the therapy, that patient will be counted as non-responder. The best overall response is the best response recorded from the start of treatment until disease progression (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The subject's best response assignment will depend on the achievement of both measurement and confirmation criteria. We will also estimate the pathological complete response rates separately for each of these tumor types. Survival and disease-free survival will be estimated using Kaplan-Meier method. With an accrual rate of 3 patients a month, we expect the study to be completed in 18 months.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Combined Modality Therapy for Esophageal Carcinoma
Number analyzed (Participants) | 55
participants | 55

2. Secondary Outcome: Evaluate Toxicity and Tolerability Including Surgical Morbidity and Mortality
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Combined Modality Therapy for Esophageal Carcinoma
Number analyzed (Participants) | 55
participants | 55

ADVERSE EVENTS:
Arm/Group | Combined Modality Therapy for Esophageal Carcinoma
Serious Adverse Events (participants affected / at risk) | 22/55
Other Adverse Events (participants affected / at risk) | 55/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined Modality Therapy for Esophageal Carcinoma (N=55)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (2)
Cardiovascular, Arrhythmia other (Cardiac disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dehydration (Gastrointestinal disorders) | 8 (10)
Diarrhea (Pts w/out col) (Gastrointestinal disorders) | 6 (6)
Dysphagia, esophagitis (Gastrointestinal disorders) | 1 (1)
Dysphagia-esophageal (Gastrointestinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Fatigue (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Neutrophil count decr (Investigations) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thrombosis (Vascular disorders) | 9 (10)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined Modality Therapy for Esophageal Carcinoma (N=55)
Alkaline phosphatase (Investigations) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (5)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Bilirubin (Investigations) | 11 (50)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Creatinine (Investigations) | 5 (30)
Diarrhea (Pts w/out col) (Gastrointestinal disorders) | 5 (5)
Dysphagia, esophagitis (Gastrointestinal disorders) | 7 (7)
Dysphagia-esophageal (Gastrointestinal disorders) | 5 (5)
Fatigue (General disorders) | 20 (20)
Hemoglobin (Hgb) (Blood and lymphatic system disorders) | 50 (200)
Hyperglycemia (Metabolism and nutrition disorders) | 36 (200)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (15)
Hypoalbuminemia (Metabolism and nutrition disorders) | 21 (40)
Hypocalcemia (Metabolism and nutrition disorders) | 44 (200)
Hypokalemia (Metabolism and nutrition disorders) | 6 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 15 (50)
Hyponatremia (Metabolism and nutrition disorders) | 5 (13)
Hypophosphatemia (Metabolism and nutrition disorders) | 40 (100)
Leukocytes (Blood and lymphatic system disorders) | 48 (250)
Lymphopenia (Blood and lymphatic system disorders) | 50 (250)
Nausea (Gastrointestinal disorders) | 11 (15)
Neutrophils/gran (Investigations) | 36 (125)
PT (Investigations) | 9 (50)
PTT (Investigations) | 10 (40)
Platelets (Investigations) | 15 (45)
SGOT (AST) (Investigations) | 5 (14)
SGPT (ALT) (Investigations) | 7 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes